CLINICAL TRIAL: NCT01739283
Title: GIP and GLP-1 in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mikkel Christensen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Mikkel Christensen, principal investigator, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-2-2009-078 33269
Record Dates: First submitted 2012-11-17; First posted 2012-12-03 (Estimated); Last update posted 2015-07-13 (Estimated); Status verified 2015-07

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Glucagon-Like Peptide 1; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hyperglycemia (Experimental): Hyperglycemic clamping
  Interventions: Other: GIP; Other: Saline
- hypoglycemia (Experimental): Hypoglycemic clamping
  Interventions: Other: GIP; Other: GLP-1; Other: Saline

INTERVENTIONS:
Other: GIP
Other: GLP-1
  Arms: hypoglycemia
Other: Saline

SUMMARY:
Investigation of Glucose-dependent Insulinotropic Polypeptide (GIP) effects at hyper and hypoglycemia in type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosed with type 1 diabetes (WHO criteria)

Exclusion Criteria:

* HbA1c > 9 %
* Liver disease (ALAT/ASAT > 2 x upper normal limit)
* Diabetic nephropathy (s-creatinine > 130 µM or albuminuria)
* Proliferative diabetic retinopathy (anamnestic)
* Severe arteriosclerosis or heart failure (NYHA group III or IV)
* Anemia
* treatment with medication not applicable to pause for 12 hours
* C-peptide increase after 50 g iv arginine

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
plasma glucagon area under curve values | approx. 15 minutes intervals, time 0 to 120 min

SECONDARY OUTCOMES:
plasma gut hormones and nutrients (absolute, incremental and area under curve values) | approx. 15 minutes intervals, time 0 to 120 min

OTHER OUTCOMES:
Glucose and glycerol tracer kinetics | approx. 15 minutes intervals, time 0 to 120 min
glucose (g/kg body weight) needed to be infuse to keep clamp | approx. 15 minutes intervals, time 0 to 120 min

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Christensen, MD, Principal Investigator — University Hospital, Gentofte, Copenhagen
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

REFERENCES:
- [Derived] Christensen M, Calanna S, Sparre-Ulrich AH, Kristensen PL, Rosenkilde MM, Faber J, Purrello F, van Hall G, Holst JJ, Vilsboll T, Knop FK. Glucose-dependent insulinotropic polypeptide augments glucagon responses to hypoglycemia in type 1 diabetes. Diabetes. 2015 Jan;64(1):72-8. doi: 10.2337/db14-0440. Epub 2014 Jul 22. PMID 25053587